CLINICAL TRIAL: NCT01558323
Title: An Open-label, Parallel-group, Single Dose Study to Assess the Pharmacokinetics of LCQ908 in Patients With Mild, Moderate and Severe Renal Impairment Compared to Age, Gender and Weight-matched Healthy Volunteers.
Brief Title: Pharmacokinetics of LCQ908 in Patients With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CLCQ908B2102
Record Dates: First submitted 2012-03-14; First posted 2012-03-20 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2014-01

CONDITIONS: Renal Impairment
Keywords: LCQ908, Renal Impairment, Pharmacokinetics
MeSH Terms: conditions — Renal Insufficiency | interventions — pradigastat

ARMS (3):
- LCQ908 (mild renal impairment plus healthy volunteers) (Experimental): Healthy subjects will be matched pair-wise by, sex, race, age (±15 years) and weight (±20%) to subjects with mild renal impairment and will receive a single 40 mg dose of LCQ908.
  Interventions: Drug: LCQ908
- LCQ908 (moderate renal impairment plus healthy volunteers) (Experimental): Healthy subjects will be matched pair-wise by, sex, race, age (±15 years) and weight (±20%) to subjects with moderate renal impairment and will receive a single 40 mg dose of LCQ908.
  Interventions: Drug: LCQ908
- LCQ908 (severe renal impairment plus healthy volunteers) (Experimental): Healthy subjects will be matched pair-wise by, sex, race, age (±15 years) and weight (±20%) to subjects with severe renal impairment and will receive a single 40 mg dose of LCQ908.
  Interventions: Drug: LCQ908

INTERVENTIONS:
Drug: LCQ908 — Participants will receive a single oral dose of LCQ908

SUMMARY:
This study will compare the pharmacokinetics of LCQ908 in subjects with varying degrees of renal impairment to healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Individuals with renal impairment only

  * Estimated Creatinine Clearance (CLcr) by the Cockroft-Gault equation ≤80mL/min;
  * Mild renal impairment defined as CLcr 50-80 mL/min
  * Moderate renal impairment defined as CLcr 30-50 mL/min
  * Severe renal impairment defined as CLcr <30 mL/min
* Healthy subjects only • Estimated CLcr by the Cockroft-Gault equation >80mL/min

Exclusion Criteria:

* All Individuals

  * A past medical history of clinically significant ECG abnormalities or a family history of a prolonged QT-interval syndrome.
  * Female subjects must be of non child bearing potential or use an effective method of contraception.
* Individuals with renal impairment

  * Renal transplant at any time.
  * Subjects undergoing any method of dialysis (hemodialysis, peritoneal dialysis) within the last 3 months.
  * History of clinically significant chronic or recurrent urinary tract infection active and requiring antibiotic treatment within the past 30 days.
  * Any medication that is contraindicated in moderate or severe renally impaired population
* Healthy subjects

  * History or presence of impaired renal function as indicated by clinically significantly abnormal creatinine or BUN and/or urea values, or abnormal urinary constituents (e.g., albuminuria)
  * Evidence of urinary obstruction or difficulty in voiding at screening
  * History or presence of hepatitis B or C and/or positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result at screening.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration (AUClast) of LCQ908 | Serial blood draws conducted on Day 1 (treatment day) followed by additional blood draws on Days 2-10,12, 14, 17, 21 and 29 post dosing
Area under the plasma concentration-time profile from time zero extrapolated to infinite time [AUC(0-inf)] of LCQ908 | Serial blood draws conducted on Day 1 (treatment day) followed by additional blood draws on Days 2-10,12, 14, 17, 21 and 29 post dosing
Maximum plasma concentration (Cmax) of LCQ908 | Serial blood draws conducted on Day 1 (treatment day) followed by additional blood draws on Days 2-10,12, 14, 17, 21 and 29 post dosing

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs), serious adverse events (SAEs) and death | Day 29
  AEs are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. SAEs are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital abnormalities or birth defects, or are other conditions which in the judgment of investigators represent significant hazards.
The apparent systemic clearance (CL/F) of LCQ908 following extra vascular administration | Serial blood draws conducted on Day 1 (treatment day) followed by additional blood draws on Days 2-10,12, 14, 17, 21 and 29 post dosing
Time to maximum plasma concentration of LCQ908 | Serial blood draws conducted on Day 1 (treatment day) followed by additional blood draws on Days 2-10,12, 14, 17, 21 and 29 post dosing
The time required for the concentration of the drug to reach half of its original value | Serial blood draws conducted on Day 1 (treatment day) followed by additional blood draws on Days 2-10,12, 14, 17, 21 and 29 post dosing
Apparent volume of distribution of LCQ908 during the terminal elimination phase following extra vascular administration | Serial blood draws conducted on Day 1 (treatment day) followed by additional blood draws on Days 2-10,12, 14, 17, 21 and 29 post dosing
LCQ908 protein binding: unbound area under curve (AUCc) of LCQ908 | 10 and 24 hours
LCQ908 protein binding: unbound observed maximum plasma (Cmax) of LCQ908 | 10 and 24 hours
LCQ908 protein binding: unbound apparent systemic clearance from plasma (CL/Fu) following extra vascular administration | 10 and 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- United States (2):
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Knoxville, Tennessee

REFERENCES:
- See also: Results for CLCQ908B2102 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=11343